CLINICAL TRIAL: NCT01811290
Title: A Single Center Prospective, Open Label, Pilot Study to Assess Change in Bone Mass Density and Select Bone Turnover Biomarkers in Gilenya Treated Versus Non-Gilenya Treated Ambulatory Subjects With a Relapsing Form of Multiple Sclerosis
Brief Title: A Pilot Study Assessing the Impact of Gilenya Therapy on Bone Density Change in Relapsing Forms of Multiple Sclerosis
Acronym: MS-BMD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Simnad, Virginia, M.D. (Individual)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Virginia I. Simnad, MD, Simnad, Virginia I. MD Medical Director, Simnad, Virginia, M.D.
Other Study IDs: MS-BMD
Record Dates: First submitted 2013-03-08; First posted 2013-03-14 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gilenya Subjects: Gilenya therapy group subjects must have been treated with Gilenya a minimum of 3 months uninterrupted prior to screening visit, and approved by the principal investigator to continue on this agent.
- Controlled Therapy Group: Control therapy group subjects must have been consistently on an FDA approved disease modifying therapy other than Gilenya or off such therapy a minimum of 6 months prior to screening visit.

SUMMARY:
The purpose of this study is to assess whether Multiple Sclerosis patients treated with Gilenya show a beneficial change over time in bone mass density and bone turnover markers as compared to matched controls treated with alternative FDA approved therapy or no therapy.

DETAILED DESCRIPTION:
To assess the effect of Gilenya on the rate of decline in bone mass density and expression of selected bone turnover biomarkers in ambulatory subject with a relapsing form of Multiple Sclerosis compared to control subjects matched for age, race, gender, duration of disease, and disability on an alternative FDA approved disease modifying therapy or no therapy at 24 months compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female subjects, 21 years of age or older.

  * Subjects must be able to give consent by signing and dating an informed consent form (written in English) prior to any study assessments being performed.
  * Ambulatory with an Expanded Disability Status Scale(EDSS) between 2.5 - 6.5 inclusive.
  * Must meet McDonald criteria for a relapsing form (relapsing remitting and secondary progressive) of Multiple Sclerosis.
  * Gilenya therapy group subjects must have been treated with Gilenya a minimum of 3 months uninterrupted prior to screening visit, and approved by the principal investigator to continue on this agent.
  * Control therapy group subjects must have been consistently on an FDA approved disease modifying therapy other than Gilenya or off such therapy a minimum of 6 months prior to screening visit.
  * Subjects must be neurologically stable and have not received any form of steroid therapy for 4 weeks prior to screening visit.
  * Subjects must abide by safety surveillance monitoring studies appropriate to their disease modifying therapy and considered standard of care. Such monitoring will be considered outside the scope of this study.
  * Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

* • Subjects must not have been treated with Fingolimod, Gilenya or other experimental Sphingosine 1-phosphate receptor agonist therapy in a clinical trial prior to enrollment in this study.

  * Subjects on an FDA approved disease modifying therapy other than Gilenya, or on no therapy, must not have received Gilenya therapy within 12 months of screening visit.
  * Current or previous use of bisphosphonate therapy, estrogen replacement, calcitonin, Depo-Provera, dehydroepiandrosterone, or methotrexate within 12 months of screening visit.
  * Medical contraindication to daily calcium intake of at least 1000 mg daily, and vitamin D3 supplementation of 800 IU daily.
  * Vitamin D insufficiency (25-hydroxy vitamin D level <=30 ng/ml) at the time of baseline visit.
  * Meeting National Osteoporosis Foundation criteria for osteoporosis requiring treatment with study prohibited therapies:
  * History of osteoporosis with baseline Dexa bone scan T score <-1.5 but >-2.0 with one or more risk factors for fracture (age >50 years, current smoking, low Body Mass Index (i.e. < 18.5), previous fragility fracture, parental history of osteoporosis or of fragility fracture of hip, femur, or vertebrae , alcohol consumption greater than 3 units per day, daily glucocorticoid usage).
  * Dexa bone scan T score < -2.0 with or without additional risk factors.
  * Subjects with Body Mass Index >=40 kg/m2 due to artifacts in Body mass density measurement with Dexa unit used.
  * Subjects with anatomical deformities or vertebral fractures that would potentially distort Body mass density measurements.
  * Current diagnosis of parathyroid disorder, untreated hyperthyroidism or hypothyroidism, renal insufficiency (Glomerular filtration rate- (GFR) <= 55), history of renal calculi or stones, uncontrolled mood disorder, drug or alcohol abuse.
  * Current use of "first generation" anticonvulsant medication (barbiturate, phenytoin, carbamazepine, valproate), or of "second generation" anticonvulsant levetiracetam (implicated recently in accelerated bone density loss). Stable use of "second generation" anticonvulsant medication (gabapentin, pregabalin, lamotrigine, topiramate, lacosamide, zonisamide, oxcarbazepine) for symptoms management will be acceptable. Stable use of dopamine reuptake inhibitor class, Serotonin Norepinephrine Reuptake Inhibitors, Selective serotonin re-uptake inhibitor antidepressant therapies will be allowed.
  * Continuous or "pulsed" treatment with a corticosteroid for any medical condition. Brief therapy with intravenous methylprednisolone 1 gram for 3-5 days with no oral taper, for a confirmed neurological relapse will be allowed.
  * Subjects must not have any unstable medical or psychiatric condition per the judgment of the principal investigator which would risk safety or completion of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 21 or older diagnosed with a relapsing form of Multiple Sclerosis. Minimum age was defined due to the limitations of site's current DXA bone scan software in scanning any person under 21 years of age. A total of 36 subjects will be recruited, with estimated 20% screen failure/early termination to allow for 30 subjects enrolled to complete the study. Racial composition of the regional population (Puget Sound of the Pacific Northwest, USA) from which study candidates will be recruited over-represents Caucasian individuals, and thus this pilot study may not be balanced for race.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assess change in bone mass density in subjects taking Gilenya versus subjects taking alternative disease modifying therapy or no therapy. | baseline and 22 months (96 weeks)
  The primary objective of this pilot study will be to assess the effect of Gilenya (fingolimod) on the rate of decline in bone mass density and expression of selected bone turnover biomarkers over 2 years in ambulatory subjects with a relapsing form of Multiple Sclerosis compared to control subjects matched for age, gender, race, duration of disease, and disability on an alternative FDA approved disease modifying therapy or no therapy.

OTHER OUTCOMES:
Interim analysis of primary outcome measures | baseline and 11 months (48 weeks)
  Assessment at week 48 of the change from baseline in bone mass density in ambulatory subjects with a relapsing form of MS treated with Gilenya compared to control subjects matched for age, gender, race, duration of disease, and disability on an alternative FDA approved disease modifying therapy or no therapy.
Interim analysis of secondary outcome measures | baseline and 11 months (48 weeks)
  expression of selected bone turnover biomarkers in ambulatory subjects with a relapsing form of Multiple Sclerosis treated with Gilenya compared to control subjects matched for age, gender, race, duration of disease, and disability on an alternative FDA approved disease modifying therapy or no therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia I Simnad, MD, Principal Investigator — Evergreen Hospital
Locations (1):
- MS Center at Evergreen Health, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No